CLINICAL TRIAL: NCT05079048
Title: Novel PEEK Retentive Elements Versus Conventional Retentive Elements in Mandibular Overdentures: A Randomized Controlled Trial
Brief Title: PEEK Retentive Elements Versus Conventional
Acronym: PEEK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sharaf Mohamed Yahia, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 19/5/2020
Record Dates: First submitted 2021-07-05; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Partially Edentulous Mandible
Keywords: Ball attachment; overdenture; patient satisfaction; PEEK; retention measurement.
MeSH Terms: conditions — Patient Satisfaction | interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional retentive element (Active Comparator): The conventional group received implant-supported mandibular overdentures retained by metal housings and nylon retentive elements,
  Interventions: Other: PEEK retentive elements
- PEEK retentive element (Experimental): PEEK group received implant-supported mandibular overdentures retained by PEEK housings ,
  Interventions: Other: PEEK retentive elements

INTERVENTIONS:
Other: PEEK retentive elements — received implant-supported mandibular overdenture retained by PEEK retentive element and housings
  Other Names: PEEK housing and clip

SUMMARY:
comparing retention and patient satisfaction of implant-supported mandibular overdentures retained by conventional nylon clip and metal housings for ball attachments versus PEEK clip and housings

DETAILED DESCRIPTION:
Background. Many patients suffer from lack of retention of conventional mandibular overdentures due to loss of clip retention over time. Computer-aided design-computer-aided manufacturing (CAD-CAM) milled polyetheretherketone PEEK materials may be used for construction of retentive housing and clip for improving retention of implant-supported overdentures.

Objective . To compare retention and patient satisfaction of implant-supported mandibular overdentures retained by conventional nylon clip and metal housings for ball attachments versus PEEK clip and housings.

Methods: Twenty-two participants were divided into 2 equal groups (n=11). The conventional group received implant-supported mandibular overdentures retained by metal housings and nylon retentive elements, while the PEEK group received implant-supported mandibular overdenture retained by PEEK retentive element and housings.The PEEK retentive elements were made by using computer-aided design and computer-aided manufacturing (CAD-CAM).Evaluation included measuring the retention by applying a gradual pulling up force by forcemeter and patient satisfaction with a 7-point visual analog scale (VAS) at overdenture insertion , 3,6, and 12 months subsequently by research interviewer.

ELIGIBILITY:
Inclusion Criteria:

* edentulous class I or II PDI classification no neuromuscular disordersand temporomandibular joint disorders

Exclusion Criteria:

* exposed to radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
retention | 3 months to six months
  measuring retention force of retentive elements using The force-meter machine (Eagle: ELT 3000) . Gradual pulling up force was applied. The record appeared at the screen of the force meter was recorded as it's single-blind measurements.

SECONDARY OUTCOMES:
patient satisfaction | 3 months to six months
  measuring patient satisfaction using Visual analog scale (VAS) was used for the evaluation of overall patient satisfaction. All questionnaires were taken by the same research interviewer (assisted interviewer) as he was blind about the type of prosthesis (double-blind) as the research interviewer is from another department

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Sharaf, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sharaf MY, Eskander A, Afify MA. Novel PEEK Retentive Elements versus Conventional Retentive Elements in Mandibular Overdentures: A Randomized Controlled Trial. Int J Dent. 2022 Feb 28;2022:6947756. doi: 10.1155/2022/6947756. eCollection 2022. PMID 35265135